CLINICAL TRIAL: NCT01513824
Title: Stress, Ongoing Self Monitoring and Ischemic Heart Disease Rehabilitation, a Randomized Controlled Trial (SongHeart)
Brief Title: Stress and Ischemic Heart Disease. The Effect of Bio Feedback Guided Stress Management on Life Quality Including Signs of Depression and Stress
Acronym: SongHeart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Jens Faber, professor, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SongHeart
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Biofeed Back Guided Stress Management; Ischemic Heart Disease
Keywords: stress; biofeed back guided treatment; acupressure; ischemic heart disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stress management, acupressure (Active Comparator): bio feedback guided stress management by daily measurement of pressure pain sensitivity followed by acupressure´for 3 months
  Interventions: Behavioral: pressure pain sensitivity measure followed bu acupressure
- bio feedback guided, stress management (No Intervention): control without treatment

INTERVENTIONS:
Behavioral: pressure pain sensitivity measure followed bu acupressure — twice daily measure of pressure pain sensitivity on the chest bone followed by stress management of which acupressure is mandatory.
  Arms: stress management, acupressure

SUMMARY:
The purpose of the study is to examine if bio feedback guided stress management by daily measurement of pressure pain sensitivity followed by acupressure reduces signs of depression and number clinical stress signs and increases quality of life in patients with stable, ischemic heart disease

DETAILED DESCRIPTION:
Primary outcome Measure:

MDI depression score (time frame 3 months) (designated as safety issue: no) The effect of 3 months twice daily measurements of Pressure Pain Sensitivity on the chest bone as a measure of the actual stress level followed by stress management of which Acupressure is mandatory

Secondary outcome measures:

1. Clinical stress signs and quality of life measures (time frame 3 months) (designated as safety issue: no) The effect of 3 months twice daily measurements of Pressure Pain Sensitivity on the chest bone as a measure of the actual stress level followed by stress management of which Acupressure is mandatory, on a Clinical Stress Signs score (56 items), SF-36 and WHO-5 questionnaires
2. Measure of Pressure Pain Sensitivity by a professional (designated as safety issue: no) The effect of 3 months twice daily measurements of pressure pain sensitivity on the chest bone as a measure of the actual stress level followed by stress management of which acupressure is mandatory
3. Measures of heart function: Blood pressure, the Pressure-Pulse Product (heart work), Heart Rate Variability inclusive response to Tilting, BNP (time frame 3 months) (designated as safety issue: no) The effect of 3 months twice daily measurements of Pressure Pain Sensitivity on the chest bone as a measure of the actual stress level followed by stress management of which Acupressure is mandatory
4. Measures of the Metabolic Syndrome: HOMA-1, Adiponectin, HBA1C, Lipids, Body Composition (time frame 3 months) (designated as safety issue: no) The effect of 3 months twice daily measurements of Pressure Pain Sensitivity on the chest bone as a measure of the actual stress level followed by stress management of which Acupressure is mandatory

Tertiary outcome Measures:

Use of health care (time frame one year after start of intervention) The effect of months twice daily measurements of Pressure Pain Sensitivity on the chest bone as a measure of the actual stress level followed by stress management of which Acupressure is mandatory, followed by 9 months bioguided feedback stress management when needed, i.e. post-study maintenance treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented stable, ischemic heart disease who have finished heart rehabilitation according to the National Guidelines > 6 months ago Actual use of aspirin, statins, and blood pressure medication according to the National Guidelines
* Age < 75 years
* Increased pressure pain sensitivity ≥60 as a sign of persistent stress

Exclusion Criteria:

* Previous diagnosed and treated psychiatric disease besides depression Other Chronic Disease with known significantly reduced life expectancy (as cancer or severe COPD)
* Other Chronic Disease with known significantly reduced Quality of Life as COPD, chronic pain conditions (but not diabetes or heart disease)
* Planned heart operation
* Changed Medication for the Heart (concerning Angina or Heart Failure) within one month
* Previous use of the Pressure Pain Sensitivity Device followed by treatment with Acupressure

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
MDI depression score | 3 months
  The effect of 3 months twice daily measurements of Pressure Pain Sensitivity on the chest bone as a measure of the actual stress level followed by stress management of which Acupressure is mandatory

SECONDARY OUTCOMES:
Clinical stress signs and quality of life measures | 3 months
  The effect of 3 months twice daily measurements of Pressure Pain Sensitivity on the chest bone as a measure of the actual stress level followed by stress management of which Acupressure is mandatory, on a Clinical Stress Signs score (56 items), SF-36 and WHO-5 questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, Herlev Hospital, Herlev, Herlev, Denmark

REFERENCES:
- [Derived] Bergmann N, Ballegaard S, Bech P, Hjalmarson A, Krogh J, Gyntelberg F, Faber J. The effect of daily self-measurement of pressure pain sensitivity followed by acupressure on depression and quality of life versus treatment as usual in ischemic heart disease: a randomized clinical trial. PLoS One. 2014 May 21;9(5):e97553. doi: 10.1371/journal.pone.0097553. eCollection 2014. PMID 24849077